CLINICAL TRIAL: NCT06724783
Title: A Randomized Controlled Clinical Trial to Compare Two Collagen Membranes for Guided Bone Regeneration (GBR) Around Dental Implants Restored with Monolithic Zirconia Single Crowns Using Three Different Veneering Designs
Brief Title: Comparison of Two Collagen Membranes for Bone Augmentation Around Dental Implants Restored with Monolithic Zirconia Single Crowns
Acronym: BioGide-Compr
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. med. dent. Malin Strasding (Other)
Responsible Party: Sponsor-Investigator, Dr. med. dent. Malin Strasding, Senior lecturer, University of Geneva, Switzerland
Organization: University of Geneva, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-D0144
Record Dates: First submitted 2024-05-15; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Tooth Extraction; Tooth Replacement
Keywords: guided bone regeneration (GBR); collagen membrane; dental implants; zirconia; monolithic ceramic fixed dental prosthesis (singe crowns)

STUDY DESIGN:
Intervention Model Description: A two parallel arm (test and control) non-inferiority, prospective, randomized controlled, monocentric, open-label clinical trial (surgical part) A three parallel arm (test, two controls) prospective, randomized controlled, monocentric, open-label clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard resorbable collagen membrane (Active Comparator): GBR with implant placement
  Interventions: Device: Collagen membrane
- Compressed, stronger resorbable collagen membrane (Experimental): GBR with implant placement
  Interventions: Device: Collagen membrane

INTERVENTIONS:
Device: Collagen membrane — Implant placement with simultaneous GBR covered with a collagen membrane

SUMMARY:
The goal of this randomized controlled clinical trial is to compare the use of two covering collagen membranes in a bone augmentation procedure around single implants and to assess three different veneering approaches on crowns in patients lacking a single tooth in the esthetic zone.

The main aims include:

1. Bone stability, i.e. the difference in the bone defect depth 4 months after bone augmentation
2. The occurrence of ceramic restoration chipping at the inserted single crowns after 5 years.

Participants will receive an implant with simultaneous bone augmentation using the bone particles and a covering collagen membrane. After the healing period, they will receive a crown restoration on the implant.

In the surgical part, researchers will compare the commonly used collagen membrane with the compressed (stronger) version of the same collagen membrane in an otherwise identical procedure to evaluate if the compressed membrane offers the same or better bone stability.

In the restorative part, researchers will compare three types of crown finishes: non-veneered, conventionally veneered and window-veneered (test group)

Participants will be asked to come to follow-up appointments over a period of 7 years. Depending on the follow-up time in the study, different dental measurements will be taken to assess the stability of the implants and restorations.

DETAILED DESCRIPTION:
Guided bone regeneration (GBR) is a standard procedure to obtain the necessary bone volume for implant placement. The most frequently performed technique relies on the application of deproteinized bone particles to augment bone volume in combination with a resorbable collagen membrane to hold the particles in place and prevent gingival connective tissue invasion. To improve the elasticity and tenacity of Bio-Gide, a new collagen membrane (compressed) has been developed and placed on the market. Potentially, improved stability of bone particles due to the more firm and rigid characteristics of the new collagen membrane would aid in better space maintenance and bone regeneration around implants.

Prosthetic restorations must be placed on implants to allow normal denture function. One of the major technical complications occurring in metal-ceramic and all-ceramic single and multiple implant-borne fixed dental prostheses (FDPs) is ceramic chipping. In highly aesthetic regions facial veneering is often necessary to overcome the aesthetic limitations of monolithic ceramic ingots. The development of a novel yet standardized approach when designing a "micro-veneered" restoration, namely window veneering, in the dental laboratory may be helpful for the reduction of chipping rates.

The primary objective of the surgery part is to determine whether the application of the new collagen membrane in a one-stage GBR+implant placement procedure results in a similar change of bone level height after 4 months compared to the application of the standard collagen membrane.

The primary objective of the restorative part is to examine the technical outcomes of the ceramic (chipping/ fracture) of three veneering designs of monolithic zirconia crowns (buccal window veneer leaving the incisal edge, standardized buccal micro-veneering or no-veneering, during 5 years of clinical function.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* ≥18 years of age
* No active periodontal disease
* Full-mouth plaque score and full-mouth bleeding score <25%.
* Patients in need of an implant-supported crown at a single-tooth gap in the aesthetic region: 11-15, 21-25, 31-35, 41-45 (FDI)
* Patients in need of GBR during implant placement (1-stage procedure)
* Presence of mesial and distal natural teeth or implant
* Implant placement at least 6 weeks after tooth extraction
* No need for soft tissue grafting

Exclusion Criteria:

* Any conditions or circumstances which would interfere with the requirements for oral surgery
* Patients with large bone defects, in need of a primary bone augmentation (two-stage procedure)
* Allergy to any implant metallic component
* Allergy to collagen
* Previous oral-maxillo-facial radiotherapy
* Any disorders in the planned implant area such as previous tumors, chronic bone
* disease (such as rheumatoid disease)
* Any ongoing application of interfering medication (steroid therapy, bisphosphonate, etc.)
* Alcohol or drug abuse
* No need for soft tissue grafting
* Patients with inadequate oral hygiene or persistent oral infection
* Clinically significant concomitant diseases (e.g. renal failure, hepatic disfunction, cardiovascular diseases)
* Heavy smokers (>10 cigarettes/day)
* Uncontrolled diabetes
* Severe bruxism or other destructive habits
* Pregnant or lactating women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Surgical part: bone stability | 4 months
  The difference in the bone defect depth after bone augmentation (baseline) and after 4 months between the groups.
Restorative part: chipping rates | 5 years
  The occurrence of ceramic chipping at the inserted single crowns

SECONDARY OUTCOMES:
Bone level changes | 1,3,5 years
  Bone width and mesial and distal bone levels
Soft tissue volume changes | 1,3,5 years
  Intraoral digital scans will be analyzed with a software to assess changes in tissue volume over time.
Restoration technical parameters | 1,3,5 years
  Prosthetic/functional and aesthetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Malin Strasding, Dr dent med, Principal Investigator — University Clinic of Dental Medicine, University of Geneva
Locations (1):
- University of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No